CLINICAL TRIAL: NCT06369883
Title: Medical Doctor, Physiatrist
Brief Title: How Often and What Type of Deformity is Detected in All Spine Radiographs?
Status: Not yet recruiting | Type: Observational
Sponsor: Bakirkoy Dr. Sadi Konuk Research and Training Hospital (Other Government)
Responsible Party: Principal Investigator, Filiz Yildiz Aydin, Medical Doctor, Bakirkoy Dr. Sadi Konuk Research and Training Hospital
Other Study IDs: 2022/41
Record Dates: First submitted 2022-08-23; First posted 2024-04-17 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Scoliosis; Kyphosis; Radiography
Keywords: scoliosis,kyphosis,radiography
MeSH Terms: conditions — Scoliosis; Kyphosis

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Subjects under 18 years of age who underwent spinal radiography: Angle measurement with Cobb method in posterior-anterior and lateral radiographs of patients who underwent spinal radiographs
  Interventions: Diagnostic Test: Spine radiography

INTERVENTIONS:
Diagnostic Test: Spine radiography — Posterior-anterior and lateral spine radiography

SUMMARY:
The study will be done retrospectively.The aim of this study is to retrospectively examine the spinal pathologies of patients with a prediagnosis of spinal deformity and for whom spinal radiography is requested and to evaluate the clinical features of these patients.

DETAILED DESCRIPTION:
Spinal radiography for scoliosis is the gold standard in the diagnosis, treatment and follow-up of spinal diseases. There are studies showing that unnecessary and repetitive radiographs of patients increase the risk of cancer in older ages. Patients should be thoroughly examined before a spine radiograph is taken. Adam's test should be applied to the patient with scoliosis findings in the physical examination. Spinal radiography for Scoliosis should be requested from those whose trunk rotation angle is 5 degrees or more during Adam's test. The diagnosis of scoliosis is made when the Cobb angle measured on posterior-anterior radiographs is greater than 10 degrees. The diagnosis of kyphosis is made when the Cobb angle measured on lateral radiographs is greater than 50 degrees. Patients with a prediagnosis of spinal deformity and spinal radiographs taken between January 2019 and September 2019 in the Radiology clinic of our hospital will be included in the study. Demographic characteristics of the patients, presence and degree of scoliosis on posterior-anterior radiographs, if present, degree of kyphosis on lateral radiographs, structural pathologies in the spine and clinical features will be investigated.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18 and under
2. Those who requested spine radiographs for scoliosis and kyphosis

Exclusion Criteria:

1. Having a history of previous spinal surgery or trauma
2. Repeated radiographs in the same patient

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients aged 18 and under, those who were requested to have spinal radiographs for scoliosis and kyphosis
Sampling Method: Probability Sample
Enrollment: 632 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-08-30 (Estimated)

PRIMARY OUTCOMES:
Who should have full spine radiographs? | 3 month
  The aim of the study is to determine the percentage of unnecessary X-rays required for he definitive diagnosis of spinal deformities and to emphasize the importance of clinical examination in requesting X-rays.

SECONDARY OUTCOMES:
We aimed to determine the frequency of kyphosis, types and percentages of scoliosis detected on the radiographs. | 3 month
  A curvature of the spine of 10° or more detected radiologically in the coronal plane is defined as scoliosis, and a curvature of over 50 degrees in the sagittal plane is defined as kyphosis. The Cobb method is calculated by measuring the angle between the parallel line drawn from the top of the top vertebra where the curvature is greatest and from the bottom of the bottom vertebra. Scoliosis is classified according to the location of the apical vertebra.

IPD SHARING:
Plan to Share IPD: Undecided